CLINICAL TRIAL: NCT00143390
Title: A Randomized, Double-Blind, Controlled Study Of Exemestane (Aromasin) Vs Anastrozole (Arimidex) As Initial Hormonal Therapy In Postmenopausal Women With Advanced/Recurrent Breast Cancer
Brief Title: Aromasin Vs Arimidex Study As Initial Hormonal Therapy In Postmenopausal Women With Advanced/Recurrent Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5991048
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2011-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: exemestane
- 2 (Experimental)
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: exemestane — take orally one tablet per day of exemestane 25 mg and one tablet per day of anastrozole placebo daily after meal
  Arms: 1
Drug: anastrozole — take orally one tablet of anastrozole 1 mg and one tablet of exemestane placebo daily after meal
  Arms: 2

SUMMARY:
To verify the non-inferiority of exemestane compared to anastrozole in time to tumor progression (TTP), the primary efficacy endpoint, in postmenopausal women with advanced/recurrent breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed breast cancer at original diagnosis. At study entry, the patient must have metastatic progressive or locally recurrent inoperable breast cancer.

Exclusion Criteria:

* Having received any hormonal therapy (e.g., Tamoxifen, LHRH-agonists) ovariectomy or any chemotherapy for advanced/recurrent breast cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2005-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- Japan (47):
  - Pfizer Investigational Site, Toyohashi, Aiche
  - Pfizer Investigational Site, Anjo, Aichi-ken
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Toyoake, Aichi-ken
  - Pfizer Investigational Site, Toyota, Aichi-ken
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Sakura, Chiba
  - Pfizer Investigational Site, Matsuyama, Ehime
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Kurume, Fukuoka
  - Pfizer Investigational Site, Kōriyama, Fukushima
  - Pfizer Investigational Site, Ōta, Gunma
  - Pfizer Investigational Site, Hiroshima, Hiroshima
  - Pfizer Investigational Site, Kure, Hiroshima
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Akashi, Hyōgo
  - Pfizer Investigational Site, Amagasaki, Hyōgo
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Higashiibaraki-gun, Ibaraki
  - Pfizer Investigational Site, Hitachi, Ibaraki
  - Pfizer Investigational Site, Morioka, Iwate
  - Pfizer Investigational Site, Kagoshima, Kagoshima-ken
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Niigata, Niigata
  - Pfizer Investigational Site, Kurashiki, Okayama-ken
  - Pfizer Investigational Site, Naha, Okinawa
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Sakai, Osaka
  - Pfizer Investigational Site, Iruma-gun, Saitama
  - Pfizer Investigational Site, Kita-adachi-gun, Saitama
  - Pfizer Investigational Site, Saitama, Saitama
  - Pfizer Investigational Site, Hamamatsu, Shizouka
  - Pfizer Investigational Site, Shizuoka, Shizuoka
  - Pfizer Investigational Site, Sunto-gun, Shizuoka
  - Pfizer Investigational Site, Shimotsuke, Tochigi
  - Pfizer Investigational Site, Utsunomiya, Tochigi
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Chuo-Ku, Tokyo
  - Pfizer Investigational Site, Koto-ku, Tokyo
  - Pfizer Investigational Site, Meguro-ku, Tokyo
  - Pfizer Investigational Site, Mitaka, Tokyo
  - Pfizer Investigational Site, Chiba

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: One tablet each of exemestane 25 mg and anastrozole placebo were orally administered once daily after a meal. The study treatment was continued until the disease progression or other discontinuation criteria were met.
- Anastrozole: One tablet each of anastrozole 1 mg and exemestane placebo were orally administered once daily after a meal. The study treatment was continued until the disease progression or other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Exemestane | Anastrozole
Started | 149 | 149
Completed | 0 | 0
Not Completed | 149 | 149
Not completed — Death | 2 | 0
Not completed — Not meeting entry criteria | 2 | 5
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Progressive disease | 119 | 115
Not completed — Protocol Violation | 2 | 0
Not completed — Study termination | 10 | 15
Not completed — Adverse Event | 9 | 8
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane | Anastrozole | Total
Number analyzed (Participants) | 149 | 149 | 298
Age, Customized [Number; unit: participants]
  18-44 years old | 2 | 0 | 2
  45-64 years old | 86 | 88 | 174
  >=65 years old | 61 | 61 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 149 | 298
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) - Expert Evaluation Committee Assessment
Description: Time in months from randomization to first documentation of objective tumor progression or death due to breast cancer, whichever comes first. Tumor progression was determined by the expert evaluation committee using RECIST version 1.0 as an at least a 20% increase in the sum of the longest diameters (SLD) of the target lesions compared to the smallest SLD since the study treatment started. For participants with bone metastasis only, at least 25% increase in the measurable lesion according to General Rules for Clinical and Pathological Study of Breast Cancer (The 14th edition).
Time Frame: Up to 2008 days of the treatment
Population: Full Analysis Set (FAS) was defined as participants who were randomized, and administered study medication at least once, and who had at least one efficacy evaluation specified in the protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 147 | 145
months | 13.8 [10.8 to 16.5] | 11.1 [10.8 to 16.6]
Statistical Analysis 1: Comparison: Exemestane vs Anastrozole; 95% Confidence Interval based on the Brookmeyer and Crowley method; Test type: Non-Inferiority or Equivalence — Non-inferiority of exemestane to anastrozole was to be concluded if the upper bound of the 95% confidence interval on the hazard ratio (exemestane/anastrozole) was ≤1.25; Hazard Ratio (HR) = 1.007, 95% CI 2-sided [0.771 to 1.317] — Disease sites, use of postoperative adjuvant antiestrogen agents therapy, and pamidronate disodium were covariates for adjustment

2. Secondary Outcome: Time to Progression (TTP) - Investigators Assessment
Description: Time in months from randomization to first documentation of objective tumor progression or death due to breast cancer, whichever comes first. Tumor progression was determined by the investigator using RECIST version 1.0 as an at least a 20% increase in the sum of the longest diameters (SLD) of the target lesions compared to the smallest SLD since the study treatment started. For participants with bone metastasis only, at least 25% increase in the measurable lesion according to General Rules for Clinical and Pathological Study of Breast Cancer (The 14th edition).
Time Frame: Up to 2008 days of the treatment
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 147 | 145
months | 13.8 [10.0 to 16.6] | 13.7 [10.9 to 16.6]
Statistical Analysis 1: Comparison: Exemestane vs Anastrozole; 95% Confidence Interval based on the Brookmeyer and Crowley method; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.059, 95% CI 2-sided [0.816 to 1.374] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Objective Response - Investigators Assessment
Description: Number of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST version 1.0). CR and PR are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as the disappearance of all target and nontarget lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters (SLD) of the targeted lesions. Objective Response (OR)= CR + PR.
Time Frame: Up to 2008 days of the treatment
Population: Full Analysis Set (FAS) was defined as participants who were randomized, and administered study medication at least once, and who had at least one efficacy evaluation specified in the protocol. Further more, participants with bone metastasis alone or not evaluable based on RECIST were excluded from this analysis.
Measure: Number; unit: participants
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 132 | 128
participants
  CR | 2 | 3
  PR | 56 | 47
  Objective Response (CR + PR) | 58 | 50

4. Secondary Outcome: Number of Participants With Clinical Benefit - Investigator Assessment
Description: Number of participants with clinical benefit based assessment of CR, PR or long-term stable disease (SD) according to the RECIST (version 1.0). CR and PR are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as the disappearance of all target and nontarget lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters (SLD) of the targeted lesions. Long-term SD was defined as SD lasted for at least 24 weeks (168 days). Clinical benefit = CR + PR + long SD
Time Frame: Up to 2008 days of the treatment
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 132 | 128
participants
  CR | 2 | 3
  PR | 56 | 47
  long-term SD | 41 | 49
  Clinical Benefit (CR+PR+long-term SD) | 99 | 99

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the date of randomization to the date of death.
Time Frame: Up to 2008 days of the treatment
Population: Full Analysis Set (FAS) was defined as subjects who were randomized, and administered study medication at least once, and who had at least one efficacy evaluation specified in the protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 147 | 145
months | NA [49.1 to NA] — OS did not reach to the median during the study. Also, the number of deaths was not sufficient to determine the upper limit of 95% confidence interval for OS. | 60.1 [48.2 to NA] — The number of deaths was not sufficient to determine the upper limit of 95% confidence interval for OS.

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from the randomization to the date of the first documentation of progressive disease (PD), symptomatic deterioration, death due to any cause, or treatment discontinuation due to adverse event, refusal or other reasons.
Time Frame: Up to 2008 days of the treatment
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 147 | 145
months | 13.6 [9.2 to 16.6] | 11.1 [9.4 to 14.1]

ADVERSE EVENTS:
Time Frame: Up to 2008 days of the treatment
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Exemestane | Anastrozole
Serious Adverse Events (participants affected / at risk) | 19/149 | 19/149
Other Adverse Events (participants affected / at risk) | 120/149 | 119/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=149) | Anastrozole (N=149)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Cataract (Eye disorders) | 2 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=149) | Anastrozole (N=149)
Constipation (Gastrointestinal disorders) | 5 | 13
Diarrhoea (Gastrointestinal disorders) | 7 | 14
Nausea (Gastrointestinal disorders) | 19 | 14
Vomiting (Gastrointestinal disorders) | 6 | 16
Fatigue (General disorders) | 10 | 6
Malaise (General disorders) | 9 | 11
Oedema peripheral (General disorders) | 6 | 12
Pyrexia (General disorders) | 11 | 15
Cystitis (Infections and infestations) | 6 | 11
Nasopharyngitis (Infections and infestations) | 54 | 55
Contusion (Injury, poisoning and procedural complications) | 5 | 8
Blood alkaline phosphatase increased (Investigations) | 12 | 11
Gamma-glutamyltransferase increased (Investigations) | 18 | 8
Weight decreased (Investigations) | 13 | 16
Weight increased (Investigations) | 12 | 7
Decreased appetite (Metabolism and nutrition disorders) | 12 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 22
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 18 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 15
Dizziness (Nervous system disorders) | 11 | 7
Headache (Nervous system disorders) | 12 | 15
Hypoaesthesia (Nervous system disorders) | 13 | 15
Insomnia (Psychiatric disorders) | 8 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Eczema (Skin and subcutaneous tissue disorders) | 4 | 9
Rash (Skin and subcutaneous tissue disorders) | 9 | 9
Hot flush (Vascular disorders) | 33 | 22
Hypertension (Vascular disorders) | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.